CLINICAL TRIAL: NCT02130193
Title: A Two Part, Phase IIa, Randomized, Placebo-controlled Study To Investigate The Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Efficacy of Oral Danirixin (GSK1325756) in Symptomatic COPD Subjects With Mild to Moderate Airflow Limitation at Risk for Exacerbations
Brief Title: Investigation of Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Efficacy of Oral Danirixin in Symptomatic COPD Subjects With Mild to Moderate Airflow Limitation at Risk for Exacerbations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200163
Record Dates: First submitted 2013-12-19; First posted 2014-05-05 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Efficacy; Danirixin; EXACT-PRO; COPD; Safety; RD; CXCR2 inhibitor; EXACT-RS; PK; HCRU exacerbations; PD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — danirixin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Subjects will receive 50 mg danirixin twice daily (BID) orally for 14 days. If the exposure to danirixin is lower than expected, after 14 days of dosing, then the dose may be increased to 75 mg BID for Part B.
  Interventions: Drug: Danirixin
- Part B (Experimental): Subjects will be randomized to receive either danirixin BID or placebo BID treatment along with standard care of treatment for 52 weeks. Subjects completing Part A and meeting the eligibility criteria for Part B could also be randomized in Part B.
  Interventions: Drug: Danirixin; Drug: Placebo

INTERVENTIONS:
Drug: Danirixin — Danirixin is available as 50 or 75 mg white, film coated immediate release tablet.
Drug: Placebo — Subjects will receive danirixin matching placebo
  Arms: Part B

SUMMARY:
The aim of this First Time in Patient study is to obtain initial information on the safety, tolerability, pharmacokinetics, pharmacodynamics and clinical efficacy of repeat daily administration of danirixin in subjects with symptomatic chronic obstructive pulmonary disease (COPD) having mild to moderate airflow limitation and are at high risk for future COPD exacerbations.

The study will be conducted in two parts. Part A will be a two week open label, single arm study in patients with COPD to obtain pharmacokinetic data and safety information of repeat dosing of danirixin in the population of interest. Approximately 10 subjects will be enrolled in Part A of the study. Progression to and dose selection for Part B will occur following review of the data collected in Part A. Part B will be a 52-week, randomized, double-blind (sponsor unblind), placebo-controlled on top of standard of care, parallel group study. Part B will evaluate several clinical efficacy assessments related to exacerbations and respiratory symptoms. Approximately 100 subjects will be enrolled with a target of 80 subjects completing 52 weeks of danirixin administration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 40 and 70 years of age inclusive, at the time of signing the informed consent
* Subjects with a documented history of COPD exacerbation(s) in the 12 months prior to study participation meeting at least one of the following criteria: >=2 COPD exacerbations resulting in prescription for antibiotics and/or oral corticosteroids or hospitalization or extended observation in a hospital emergency room or outpatient center; 1 COPD exacerbation resulting in prescription for antibiotics and/or oral corticosteroids or hospitalization or extended observation in a hospital emergency room or outpatient center and a plasma fibrinogen concentration at screening >=3.5 milligram/milliliter (mg/mL)
* Diagnosis of symptomatic chronic obstructive pulmonary disease with mild to moderate airflow obstruction (COPD-GOLD I or II) for at least 2 years based on American Thoracic Society (ATS)/ European Respiratory Society (ERS) current guidelines or symptoms consistent with COPD for at least 2 years
* Subjects with a post-bronchodilator FEV1/FVC ratio of < 0.7 and FEV1 >=50% of predicted normal value calculated using National Health and Nutrition Examination Survey (NHANES) III reference equation at Visit 1
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli international units/mL (MIU/mL) and estradiol < 40 picogram (pg)/mL (<147 picomole/Liter [pmol/L]) is confirmatory]. Females on hormone replacement therapy (HRT) will not be enrolled in the study.
* Body weight >=45 kilogram (kg)
* Current smokers and former smokers with a cigarette smoking history of >=10 pack years (1 pack year =20 cigarettes smoked per day for 1 year or equivalent). Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1
* Subjects with a history of respiratory symptoms, including chronic cough and/or mucus hypersecretion on most days for at least the previous 3 months prior to Visit 1
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) <2x upper limit of normal (ULN); alkaline phosphatase and bilirubin <=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Able to perform lung function tests reliably
* Based on single or averaged corrected QT (QTc) values of triplicate ECGs obtained over a brief recording period: Fridericia-corrected QTc (QTcF) < 450 milliseconds (msec); or QTc < 480 msec in subjects with Bundle Branch Block
* Subjects must have the ability to use an electronic diary on a daily basis [Part B only]
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* Diagnosis of asthma, or other clinically relevant lung disease (other than COPD), e.g. sarcoidosis, tuberculosis, pulmonary fibrosis, severe bronchiectasis or lung cancer; Subject with alpha-1-antitrypsin deficiency as the underlying cause of COPD
* Pulse Oximetry levels <88% (at rest on room air) at screening
* Less than 14 days have elapsed from completion of a course of antibiotics or oral corticosteroids for a recent COPD exacerbation.
* Diagnosis of Pneumonia (chest X-Ray or computed tomography [CT] confirmed) within the last 3 months prior to screening
* History or current evidence of clinically significant renal disease, diabetes mellitus/metabolic syndrome, hypertension or any other clinically significant cardiovascular, neurological, endocrine, or hematological abnormalities that are uncontrolled on permitted therapy. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subjects at risk through study participation, or which would affect the safety analysis or other analysis if the disease/condition exacerbated during the study.
* A positive pre-study drug/alcohol screen
* A positive test for human immunodeficiency virus (HIV) antibody
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: For non United States of America (US) sites: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits; For US sites: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Current or expected use of proton pump inhibitors or histamine H2-receptor antagonists during the study period
* Chest X-ray (posteroanterior with lateral) or CT scan reveals evidence of pneumonia or a clinically significant abnormality not believed to be due to the presence of COPD (historic data up to 1 yr may be used).
* Subjects with peripheral blood neutrophil count (PBN) <2x10^9/Liter
* Subject with history of previous lung surgery (e.g. lobectomy, pneumonectomy, or lung volume reduction)
* Requiring the use of oral or injectable Cytochrome P450 3A4 (CYP3A4) or breast cancer resistance protein (BCRP) substrates with a narrow therapeutic index

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-02-13 (Actual); Primary Completion 2016-08-29 (Actual); Study Completion 2016-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- United States (6):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Oaks, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Spartanburg, South Carolina
- Germany (8):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin

REFERENCES:
- [Derived] Lazaar AL, Miller BE, Tabberer M, Yonchuk J, Leidy N, Ambery C, Bloomer J, Watz H, Tal-Singer R. Effect of the CXCR2 antagonist danirixin on symptoms and health status in COPD. Eur Respir J. 2018 Oct 4;52(4):1801020. doi: 10.1183/13993003.01020-2018. Print 2018 Oct. No abstract available. PMID 30139779

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2 part study. In Part A, an open label, single arm, participants (par.) received danrixin 50 milligrams (mg) twice daily (BID) for 2 weeks. In Part B, a randomized (1:1), double-blind (sponsor unblinded) placebo controlled on top of standard of care study, par. received DNX 75 mg BID in one arm and placebo in the other arm for 52 weeks.
Pre-assignment Details: A total of 19 par. in Part A were screened (10 failed) and 9 were randomized in a 2-week treatment period (TP) followed by a follow-up visit (FU) at 7- 14 days after last dose. A total of 127 par. in Part B were screened (34 failed) and 93 were randomized in a 52-week TP followed by a FU at 14- 28 days after last dose of the study.
Groups:
- Part A: 4-week Open-label Period: DNX 50 mg: Participants received one immediate release tablet of danirixin (DNX) 50 mg BID with food and water for 2 weeks. Participants were permitted to continue taking inhaled maintenance medications. Rescue medications for acute symptoms were also permitted (e.g. short acting bronchodilators).
- Part B: 52-week Double-blind Period: Placebo: Participants received one tablet of placebo twice daily with food and water for 52 weeks. It was administered on top of the participant's current standard of care. Participants were permitted to continue taking inhaled maintenance medications. Rescue medications for acute symptoms were also permitted (e.g. short acting bronchodilators).
- Part B: 52-week Double-blind Period: DNX 75 mg: Participants received one immediate release tablet of danirixin (DNX) 75 mg BID with food and water for 52 weeks. It was administered on top of the participant's current standard of care. Participants were permitted to continue taking inhaled maintenance medications. Rescue medications for acute symptoms were also permitted (e.g. short acting bronchodilators).
Period: Part A: 4-week Open-label Period
Arm/Group | Part A: 4-week Open-label Period: DNX 50 mg | Part B: 52-week Double-blind Period: Placebo | Part B: 52-week Double-blind Period: DNX 75 mg
Started | 9 | 0 | 0
Completed | 9 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part B: 52-week Double-blind Period
Arm/Group | Part A: 4-week Open-label Period: DNX 50 mg | Part B: 52-week Double-blind Period: Placebo | Part B: 52-week Double-blind Period: DNX 75 mg
Started | 0 | 48 | 45
Completed | 0 | 38 | 37
Not Completed | 0 | 10 | 8
Not completed — Adverse Event | 0 | 5 | 3
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Data for Part B is presented.
Groups:
- Placebo: Participants received one tablet of placebo twice daily with food and water for 52 weeks. It was administered on top of the participant's current standard of care. Participants were permitted to continue taking inhaled maintenance medications. Rescue medications for acute symptoms were also permitted (e.g. short acting bronchodilators).
- DNX 75 mg: Participants received one immediate release tablet of danirixin (DNX) 75 mg BID with food and water for 52 weeks. It was administered on top of the participant's current standard of care. Participants were permitted to continue taking inhaled maintenance medications. Rescue medications for acute symptoms were also permitted (e.g. short acting bronchodilators).
- Total: Total of all reporting groups
Arm/Group | Placebo | DNX 75 mg | Total
Number analyzed (Participants) | 48 | 45 | 93
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.8 (7.32) | 62.4 (6.91) | 60.5 (7.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 23 | 22 | 45
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 47 | 45 | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) and, Serious Adverse Event (SAE) in Part A
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention, events associated with liver injury and impaired liver function were categorized as SAE. Participants with any AE or SAE were summarized. Participants with AE or SAE occurrences >= 5 percent were summarized. All Subjects Population comprised of all participants who were screened and for whom a record existed on the study database.
Time Frame: Up to Day 28 in Part A
Population: All Subjects Population
Measure: Number; unit: Participants
Groups:
- DNX 50 mg: Participants received one immediate release tablet of danirixin (DNX) 50 mg BID with food and water for 2 weeks. Participants were permitted to continue taking inhaled maintenance medications. Rescue medications for acute symptoms were also permitted (e.g. short acting bronchodilators).
Arm/Group | DNX 50 mg
Number analyzed (Participants) | 9
Participants
  AE | 5
  SAEs | 1

2. Primary Outcome: Number of Participants With Any AE and SAE in Part B
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention, events associated with liver injury and impaired liver function were categorized as SAE. Participants with AE or SAE occurrences >= 5 percent were summarized.
Time Frame: Up to Day 392 in Part B
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
Participants
  AE | 25 | 25
  SAEs | 10 | 10

3. Primary Outcome: Number of Participants With Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), Pulse Rate, Respiratory Rate and Body Temperature Abnormalities of Potential Clinical Importance in Part A
Description: Vital signs including SBP, DBP, pulse rate, respiratory rate and body temperature were taken on Day 1 pre-dose and on Day 14 and at Follow-up (Day 21 to 28) in Part A. Measurements were obtained in a semi-supine/ supine position after 5 minutes rest. The mean of replicate assessments at any given time point was used as the value for that time point. SBP <90 or >160 millimeter of mercury (mmHg); DBP <40 or >110 mmHg, pulse rate <35 or >120 beats per minute (bpm) and respiratory rate <8 or >30 breaths per minute were considered as values of potential clinical importance and were presented as 'High' or 'Low' values. Intent-to-Treat (ITT) Population comprised of all randomized par. who received at least one dose of study medication.
Time Frame: Up to Day 28 in Part A
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | DNX 50 mg
Number analyzed (Participants) | 9
Participants
  SBP, Day 14, low | 0
  SBP, Day 14, high | 2
  DBP, Day 14, low | 0
  DBP, Day 14, high | 1

4. Primary Outcome: Number of Participants With Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), Pulse Rate and Respiratory Rate Abnormalities of Potential Clinical Importance in Part B
Description: Vital signs including SBP, DBP, pulse rate and respiratory rate were taken on Day 1 pre-dose and on Day 28, 56, 112, 168, 280, 364 and at Follow-up (Day 378 to 392) in Part B. Measurements were obtained in a semi-supine/ supine position after 5 minutes rest. The mean of replicate assessments at any given time point was used as the value for that time point. SBP <90 or >160 mmHg, DBP <40 or >110 mmHg, pulse rate <35 or >120 bpm and respiratory rate <8 or >30 breaths per minute were considered as values of potential clinical importance and were presented as 'High' or 'Low' values. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
Participants
  SBP, Day 1, low, n=48, 45 | 0 | 0
  SBP, Day 1, high, n=48, 45 | 0 | 2
  SBP, Day 28, low, n=47, 44 | 0 | 0
  SBP, Day 28, high, n=47, 44 | 0 | 3
  SBP, Day 56, low, n=46, 41 | 0 | 0
  SBP, Day 56, high, n=46, 41 | 2 | 2
  SBP, Day 112, low, n=46, 40 | 0 | 0
  SBP, Day 112, high, n=46, 40 | 3 | 2
  SBP, Day 168, low, n=44, 39 | 0 | 0
  SBP, Day 168, high, n=44, 39 | 2 | 3
  SBP, Day 280, low, n=39, 37 | 1 | 0
  SBP, Day 280, high, n=39, 37 | 2 | 2
  SBP, Day 364, low, n=39, 37 | 0 | 0
  SBP, Day 364, high, n=39, 37 | 1 | 4
  DBP, Day 280, low, n=39, 37 | 0 | 0
  DBP, Day 280, high, n=39, 37 | 1 | 0
  Respiratory rate, Day 1, low, n=48, 45 | 1 | 0
  Respiratory rate, Day 1, high, n=48, 45 | 1 | 0
  Respiratory rate, Day 56, low, n=46, 41 | 0 | 0
  Respiratory rate, Day 56, high, n=46, 41 | 2 | 0
  Respiratory rate, Day 112, low, n=46, 40 | 1 | 0
  Respiratory rate, Day 112, high, n=46, 40 | 0 | 0
  Respiratory rate, Day 168, low, n=44, 39 | 0 | 0
  Respiratory rate, Day 168, high, n=44, 39 | 0 | 1

5. Primary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) in Part A
Description: 12-lead ECG was taken on Day 1 pre-dose and on Follow-up visit (Day 21 to 28) in Part A using an ECG machine. Triplicate reading were taken on Day 1 pre-dose. Participants with abnormal-clinically not significant (NCS) and abnormal-clinically significant (CS) findings were sumarized.
Time Frame: Up to Day 28 in Part A
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | DNX 50 mg
Number analyzed (Participants) | 9
Participants
  Abnormal-NCS, Day 1, pre-dose | 3
  Abnormal-CS, Day 1, pre-dose | 0
  Abnormal-NCS, Day 1, pre-dose 2 | 2
  Abnormal-CS, Day 1, pre-dose 2 | 0
  Abnormal-NCS, Day 1, pre-dose 3 | 2
  Abnormal-CS, Day 1, pre-dose 3 | 0

6. Primary Outcome: Number of Participants With Abnormal 12-lead ECG in Part B
Description: 12-lead ECG was taken on Day 1 pre-dose and on Day 28, 168 and at Follow-up (Day 378 to 392) in Part B using an ECG machine. Participants with abnormal-NCS and abnormal-CS findings were sumarized. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
Participants
  Abnormal-NCS, Day 28, n=47, 44 | 20 | 16
  Abnormal-CS, Day 28, n=47, 44 | 0 | 1
  Abnormal-NCS, Day 168, n=44, 38 | 15 | 11
  Abnormal-CS, Day 168, n=44, 38 | 0 | 0

7. Primary Outcome: Number of Participants With Hematology Values of Potential Clinical Importance in Part A
Description: Blood samples were collected at Screening and Day 14 in Part A to evaluate hematology parameters which included hemoglobin, hematocrit, basophils, eosinophils, lymphocytes, monocytes, neutrophils, mean corpuscular hemoglobin concentration (MCHC), mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), red blood cell (RBC) count, white blood cell (WBC) count, platelet count and reticulocyte count. Hematology values of potential clinical importance were presented as 'High' or 'Low' values based on the reference laboratory standards.
Time Frame: Up to Day 28 in Part A
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | DNX 50 mg
Number analyzed (Participants) | 9
Participants
  RBC count, Day 14, low | 1
  Category title 2. RBC count, Day 14, high | 0

8. Primary Outcome: Number of Participants With Hematology Values of Potential Clinical Importance in Part B
Description: Blood samples were collected at Screening and on Day 28, 168, and 364 in Part B to evaluate hematology parameters which included hemoglobin, hematocrit, basophils, eosinophils, lymphocytes, monocytes, neutrophils, MCHC, MCH, MCV, RBC count, WBC count, platelet count and reticulocyte count. Hematology values of potential clinical importance were presented as 'High' or 'Low' values based on the reference laboratory standards. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
Participants
  Platelet count, Day 28, low, n=46, 43 | 0 | 1
  Platelet count, Day 28, high, n=46, 43 | 0 | 0
  RBC count, Day 28, low, n=46, 43 | 0 | 1
  RBC count, Day 28, high, n=46, 43 | 0 | 0
  Platelet count, Day 168, low, n=43, 38 | 0 | 1
  Platelet count, Day 168, high, n=43, 38 | 1 | 0
  RBC count, Day 168, low, n=44, 38 | 2 | 1
  RBC count, Day 168, high, n=44, 38 | 0 | 0
  WBC count, Day 168, low, n=44, 38 | 0 | 0
  WBC count, Day 168, high, n=44, 38 | 1 | 0
  Platelet count, Day 364, low, n=39, 36 | 0 | 1
  Platelet count, Day 364, high, n=39, 36 | 0 | 0
  RBC count, Day 364, low, n=39, 36 | 2 | 1
  RBC count, Day 364, high, n=39, 36 | 0 | 0

9. Primary Outcome: Number of Participants With Clinical Chemistry Values of Potential Clinical Importance in Part A
Description: Blood samples were collected at Screening and Day 14 in Part A to evaluate clinical chemistry parameters which included alanine aminotransferase (ALT), albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), total bilirubin, calcium, bicarbonate, chloride, creatinine, direct bilirubin, gamma glutamyl transferase (GGT), glucose, potassium, total protein, sodium, blood urea nitrogen (BUN) and uric acid. Additional liver monitoring chemistry (ALT, AST, ALP and total and direct bilirubin) was done on Day 1 pre-dose. Clinical chemistry values of potential clinical importance were presented as 'High' or 'Low' values based on the reference laboratory standards.
Time Frame: Up to Day 28 in Part A
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | DNX 50 mg
Number analyzed (Participants) | 9
Participants
  GGT, Day 14, low | 0
  GGT, Day 14, high | 2
  Uric acid, Day 14, low | 0
  Uric acid, Day 14, high | 8

10. Primary Outcome: Number of Participants With Clinical Chemistry Values of Potential Clinical Importance in Part B
Description: Blood samples were collected at Screening and on Day 28, 168 and 364 in Part B to evaluate clinical chemistry parameters which included ALT, albumin, ALP, AST, total bilirubin, calcium, bicarbonate, chloride, creatinine, direct bilirubin, GGT, glucose, potassium, total protein, sodium, BUN and uric acid. Clinical chemistry values of potential clinical importance were presented as 'High' or 'Low' values based on the reference laboratory standards. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
Participants
  Creatinine, Day 28, low, n=47, 44 | 0 | 0
  Creatinine, Day 28, high, n=47, 44 | 0 | 1
  GGT, Day 28, low, n=47, 44 | 0 | 0
  GGT, Day 28, high, n=47, 44 | 7 | 3
  Uric acid, Day 28, low, n=47, 44 | 0 | 0
  Uric acid, Day 28, high, n=47, 44 | 47 | 44
  ALP, Day 84, low, n=46, 40 | 0 | 0
  ALP, Day 84, high, n=46, 40 | 0 | 1
  ALT, Day 84, low, n=46, 40 | 0 | 0
  ALT, Day 84, high, n=46, 40 | 0 | 1
  AST, Day 84, low, n=46, 40 | 0 | 0
  AST, Day 84, high, n=46, 40 | 0 | 1
  GGT, Day 168, low, n=43, 39 | 0 | 0
  GGT, Day 168, high, n=43, 39 | 5 | 1
  Uric acid, Day 168, low, n=43, 39 | 0 | 0
  Uric acid, Day 168, high, n=43, 39 | 43 | 39
  Direct bilirubin, Day 364, low, n=39, 37 | 0 | 0
  Direct bilirubin, Day 364, high, n=39, 37 | 1 | 0
  Total bilirubin, Day 364, low, n=39, 37 | 0 | 0
  Total bilirubin, Day 364, high, n=39, 37 | 1 | 0
  GGT, Day 364, low, n=39, 37 | 0 | 0
  GGT, Day 364, high, n=39, 37 | 5 | 1
  Uric acid, Day 364, low, n=39, 37 | 0 | 0
  Uric acid, Day 364, high, n=39, 37 | 39 | 37

11. Primary Outcome: Number of Participants With Urinalysis Dipstick Results in Part A
Description: Test strip urinalysis was done for glucose, ketones, occult blood and protein at Screening and Day 14 in Part A. Results were presented as negative, trace, 1+, 2+ and 3+ for glucose, ketones, occult blood and protein. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Day 28 in Part A
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | DNX 50 mg
Number analyzed (Participants) | 9
Participants
  Occult blood, Day 14, negative, n=9 | 9
  Glucose, Day 14, negative, n=9 | 9
  Ketones, Day 14, negative, n=9 | 9
  Protein, Day 14, 1+, n=9 | 1
  Protein, Day 14, negative, n=9 | 8
  Urine microscopy-RBC, Day 14, not seen, n=1 | 1
  Urine microscopy-WBC, Day 14, not seen, n=1 | 1

12. Primary Outcome: Number of Participants With Urinalysis Dipstick Results in Part B
Description: Test strip urinalysis was done for glucose, ketones, occult blood and protein at Screening and on Day 28, 168, 224 and 364 in Part B. Results were presented as negative, trace, 1+, 2+ and 3+ for glucose, ketones, occult blood and protein. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
Participants
  Occult blood, Day 28, trace, n=47, 44 | 0 | 2
  Occult blood, Day 28, 1+, n=47, 44 | 3 | 0
  Occult blood, Day 28, negative, n=47, 44 | 44 | 42
  Glucose, Day 28, trace, n=47, 44 | 0 | 1
  Glucose, Day 28, 1+, n=47, 44 | 1 | 0
  Glucose, Day 28, 3+, n=47, 44 | 0 | 2
  Glucose, Day 28, negative, n=47, 44 | 46 | 41
  Ketones, Day 28, trace, n=47, 44 | 3 | 2
  Ketones, Day 28, negative, n=47, 44 | 44 | 42
  Protein, Day 28, trace, n=47, 44 | 2 | 1
  Protein, Day 28, 1+, n=47, 44 | 2 | 2
  Protein, Day 28, negative, n=47, 44 | 43 | 41
  Occult blood, Day 168, trace, n=42, 36 | 3 | 2
  Occult blood, Day 168, 1+, n=42, 36 | 1 | 1
  Occult blood, Day 168, 3+, n=42, 36 | 1 | 0
  Occult blood, Day 168, negative, n=42, 36 | 37 | 33
  Glucose, Day 168, 2+, n=42, 36 | 1 | 0
  Glucose, Day 168, negative, n=42, 36 | 41 | 36
  Ketones, Day 168, trace, n=42, 36 | 3 | 0
  Ketones, Day 168, negative, n=42, 36 | 39 | 36
  Protein, Day 168, trace, n=42, 36 | 2 | 1
  Protein, Day 168, 1+, n=42, 36 | 1 | 2
  Protein, Day 168, 2+, n=42, 36 | 1 | 0
  Protein, Day 168, negative, n=42, 36 | 38 | 33
  Occult blood, Day 224, negative, n=1, 0 | 1 | 0
  Glucose, Day 224, negative, n=1, 0 | 1 | 0
  Ketones, Day 224, negative, n=1, 0 | 1 | 0
  Protein, Day 224, negative, n=1, 0 | 1 | 0
  Occult blood, Day 364, trace, n=38, 36 | 3 | 2
  Occult blood, Day 364, 1+, n=38, 36 | 2 | 1
  Occult blood, Day 364, negative, n=38, 36 | 33 | 33
  Glucose, Day 364, trace, n=38, 36 | 1 | 0
  Glucose, Day 364, 2+, n=38, 36 | 1 | 0
  Glucose, Day 364, negative, n=38, 36 | 36 | 36
  Ketones, Day 364, trace, n=38, 36 | 3 | 0
  Ketones, Day 364, negative, n=38, 36 | 35 | 36
  Protein, Day 364, trace, n=38, 36 | 3 | 0
  Protein, Day 364, 1+, n=38, 36 | 1 | 2
  Protein, Day 364, 2+, n=38, 36 | 1 | 1
  Protein, Day 364, negative, n=38, 36 | 33 | 33

13. Primary Outcome: Change From Baseline in Urine Power of Hydrogen (pH) at Day 14 in Part A
Description: Urinalysis including urine pH was done at Screening and Day 14 in Part A. Baseline was considered as the measurement obtained at Screening (Day -1). The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Up to Day 28 in Part A
Population: ITT Population
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | DNX 50 mg
Number analyzed (Participants) | 9
pH | -0.06 (1.488)

14. Primary Outcome: Change From Baseline in Urine pH in Part B
Description: Urinalysis including urine pH was done at Screening and on Day 28, 168 and 364 in Part B. Baseline was considered as the measurement obtained at Screening (Day -1). The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
pH
  Day 28, n=45, 43 | -0.17 (0.648) | -0.10 (0.552)
  Day 168, n=40, 35 | -0.18 (0.694) | -0.13 (0.751)
  Day 364, n=36, 35 | -0.29 (0.731) | -0.07 (0.768)

15. Primary Outcome: Change From Baseline in Urine Specific Gravity of Urine in Part A
Description: Urinalysis including urine specific gravity was done at Screening and Day 14 in Part A. Baseline was considered as the measurement obtained at Screening (Day -1). The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Up to Day 28 in Part A
Population: ITT Population
Measure: Mean (Standard Deviation); unit: urine specific gravity
Arm/Group | DNX 50 mg
Number analyzed (Participants) | 9
urine specific gravity | -0.0008 (0.00817)

16. Primary Outcome: Change From Baseline in Urine Specific Gravity of Urine in Part B
Description: Urinalysis including urine specific gravity was done at Screening and on Day 28, 168 and 364 in Part B. Baseline was considered as the measurement obtained at Screening (Day -1). The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Mean (Standard Deviation); unit: urine specific gravity
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
urine specific gravity
  Day 28, n=45, 43 | -0.0011 (0.00643) | -0.0008 (0.00536)
  Day 168, n=40, 35 | -0.0012 (0.00771) | -0.0002 (0.00748)
  Day 364, n=36, 35 | 0.0004 (0.00569) | 0.0013 (0.00561)

17. Primary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) and Forced Vital Capacity (FVC) at the Indicated Time Points in Part A
Description: FEV1 measures how much air a person can exhale during a forced breath in 1 second. FVC is the total amount of air exhaled during the FEV test. FEV1 and FVC were performed at Screening and on Day 1, 14 and at Follow-up visit (Day 21 to 28). FEV1 and FVC assessments at each time point (post-bronchodilator) were taken in triplicate. The maximum of the triplicate assessments were used. Baseline was considered as the measurement obtained at Day 1 pre-dose. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Up to Day 28 in Part A
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | DNX 50 mg
Number analyzed (Participants) | 9
Liter
  FEV1, Day 14 | 0.0978 (0.10378)
  FVC, Day 14 | 0.2233 (0.25407)

18. Primary Outcome: Change From Baseline in FEV1 and FVC at the Indicated Time Points in Part B
Description: FEV1 and FVC were performed at Screening and on Day 1, 28, 56, 112, 168, 280, 364 and at Follow-up (Day 378 to 392) in Part B. FEV1 and FVC assessments at each time point (post-bronchodilator) were taken in triplicate. The maximum of the triplicate assessments were used. Baseline was considered as the measurement obtained at Day 1 pre-dose. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Statistical analysis was performed using a repeated measures mixed effects model in a Bayesian framework. The estimate of the treatment difference and corresponding 95 percent credible interval was constructed for the difference between danirixin and placebo for each visit. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
Liter
  FEV1, Day 28, n=47, 44 | -0.018 (0.2049) | 0.048 (0.1433)
  FEV1, Day 56, n=46, 41 | 0.048 (0.3377) | 0.017 (0.1633)
  FEV1, Day 112, n=45, 39 | 0.011 (0.2431) | 0.088 (0.3044)
  FEV1, Day 168, n=44, 39 | 0.018 (0.2944) | 0.015 (0.2129)
  FEV1, Day 280, n=39, 37 | -0.012 (0.3300) | 0.043 (0.2310)
  FEV1, Day 364, n=39, 37 | -0.009 (0.2746) | 0.028 (0.2988)
  FVC, Day 28, n=47, 44 | 0.027 (0.3407) | 0.022 (0.2845)
  FVC, Day 56, n=46, 41 | 0.046 (0.4344) | 0.036 (0.2706)
  FVC, Day 112, n=45, 39 | 0.024 (0.4195) | 0.014 (0.3714)
  FVC, Day 168, n=44, 39 | -0.061 (0.3956) | -0.005 (0.3301)
  FVC, Day 280, n=39, 37 | -0.020 (0.5966) | 0.041 (0.4271)
  FVC, Day 364, n=39, 37 | -0.021 (0.4290) | 0.008 (0.4190)
Statistical Analysis 1: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.87, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.06, 95% CI 2-sided [-0.05 to 0.18], Standard Deviation 0.06 — FEV1, Day 28. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 2: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.78, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.02 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.06, 95% CI 2-sided [-0.05 to 0.18], Standard Deviation 0.06 — FEV1, Day 28. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 3: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.67, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.04 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.06, 95% CI 2-sided [-0.05 to 0.18], Standard Deviation 0.06 — FEV1, Day 28. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 4: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.52, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.06 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.06, 95% CI 2-sided [-0.05 to 0.18], Standard Deviation 0.06 — FEV1, Day 28. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 5: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.39, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.08 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.06, 95% CI 2-sided [-0.05 to 0.18], Standard Deviation 0.06 — FEV1, Day 28. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 6: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.26, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.10 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.06, 95% CI 2-sided [-0.05 to 0.18], Standard Deviation 0.06 — FEV1, Day 28. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 7: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.31, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.04, 95% CI 2-sided [-0.20 to 0.09], Standard Deviation 0.07 — FEV1, Day 56. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 8: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.22, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.02 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.04, 95% CI 2-sided [-0.20 to 0.09], Standard Deviation 0.07 — FEV1, Day 56. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 9: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.14, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.04 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.04, 95% CI 2-sided [-0.20 to 0.09], Standard Deviation 0.07 — FEV1, Day 56. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 10: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.09, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.06 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.04, 95% CI 2-sided [-0.20 to 0.09], Standard Deviation 0.07 — FEV1, Day 56. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 11: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.05, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.08 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.04, 95% CI 2-sided [-0.20 to 0.09], Standard Deviation 0.07 — FEV1, Day 56. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 12: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.03, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.10 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.04, 95% CI 2-sided [-0.20 to 0.09], Standard Deviation 0.07 — FEV1, Day 56. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 13: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.85, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.08, 95% CI 2-sided [-0.06 to 0.23], Standard Deviation 0.08 — FEV1, Day 112. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 14: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.79, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.02 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.08, 95% CI 2-sided [-0.06 to 0.23], Standard Deviation 0.08 — FEV1, Day 112. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 15: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.71, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.04 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.08, 95% CI 2-sided [-0.06 to 0.23], Standard Deviation 0.08 — FEV1, Day 112. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 16: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.61, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.06 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.08, 95% CI 2-sided [-0.06 to 0.23], Standard Deviation 0.08 — FEV1, Day 112. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 17: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.51, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.08 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.08, 95% CI 2-sided [-0.06 to 0.23], Standard Deviation 0.08 — FEV1, Day 112. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 18: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.41, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.10 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.08, 95% CI 2-sided [-0.06 to 0.23], Standard Deviation 0.08 — FEV1, Day 112. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 19: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.47, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.00, 95% CI 2-sided [-0.16 to 0.14], Standard Deviation 0.07 — FEV1, Day 168. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 20: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.36, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.02 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.00, 95% CI 2-sided [-0.16 to 0.14], Standard Deviation 0.07 — FEV1, Day 168. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 21: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.26, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.04 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.00, 95% CI 2-sided [-0.16 to 0.14], Standard Deviation 0.07 — FEV1, Day 168. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 22: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.19, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.06 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.00, 95% CI 2-sided [-0.16 to 0.14], Standard Deviation 0.07 — FEV1, Day 168. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 23: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.13, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.08 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.00, 95% CI 2-sided [-0.16 to 0.14], Standard Deviation 0.07 — FEV1, Day 168. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 24: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.09, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.10 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.00, 95% CI 2-sided [-0.16 to 0.14], Standard Deviation 0.07 — FEV1, Day 168. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 25: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.78, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.06, 95% CI 2-sided [-0.11 to 0.20], Standard Deviation 0.08 — FEV1, Day 280. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 26: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.69, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.02 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.06, 95% CI 2-sided [-0.11 to 0.20], Standard Deviation 0.08 — FEV1, Day 280. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 27: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.59, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.04 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.06, 95% CI 2-sided [-0.11 to 0.20], Standard Deviation 0.08 — FEV1, Day 280. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 28: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.50, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.06 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.06, 95% CI 2-sided [-0.11 to 0.20], Standard Deviation 0.08 — FEV1, Day 280. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 29: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.39, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.08 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.06, 95% CI 2-sided [-0.11 to 0.20], Standard Deviation 0.08 — FEV1, Day 280. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 30: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.30, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.10 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.06, 95% CI 2-sided [-0.11 to 0.20], Standard Deviation 0.08 — FEV1, Day 280. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 31: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.68, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.04, 95% CI 2-sided [-0.14 to 0.20], Standard Deviation 0.08 — FEV1, Day 364. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 32: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.59, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.02 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.04, 95% CI 2-sided [-0.14 to 0.20], Standard Deviation 0.08 — FEV1, Day 364. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 33: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.50, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.04 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.04, 95% CI 2-sided [-0.14 to 0.20], Standard Deviation 0.08 — FEV1, Day 364. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 34: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.40, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.06 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.04, 95% CI 2-sided [-0.14 to 0.20], Standard Deviation 0.08 — FEV1, Day 364. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 35: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.30, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.08 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.04, 95% CI 2-sided [-0.14 to 0.20], Standard Deviation 0.08 — FEV1, Day 364. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 36: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.22, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.10 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.04, 95% CI 2-sided [-0.14 to 0.20], Standard Deviation 0.08 — FEV1, Day 364. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 37: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.41, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.02, 95% CI 2-sided [-0.19 to 0.13], Standard Deviation 0.08 — FVC, Day 28. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 38: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.32, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.02 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.02, 95% CI 2-sided [-0.19 to 0.13], Standard Deviation 0.08 — FVC, Day 28. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 39: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.24, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.04 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.02, 95% CI 2-sided [-0.19 to 0.13], Standard Deviation 0.08 — FVC, Day 28. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 40: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.16, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.06 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.02, 95% CI 2-sided [-0.19 to 0.13], Standard Deviation 0.08 — FVC, Day 28. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 41: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.11, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.08 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.02, 95% CI 2-sided [-0.19 to 0.13], Standard Deviation 0.08 — FVC, Day 28. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 42: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.07, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.10 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.02, 95% CI 2-sided [-0.19 to 0.13], Standard Deviation 0.08 — FVC, Day 28. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 43: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.41, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.02, 95% CI 2-sided [-0.20 to 0.15], Standard Deviation 0.09 — FVC, Day 56. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 44: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.32, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.02 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.02, 95% CI 2-sided [-0.20 to 0.15], Standard Deviation 0.09 — FVC, Day 56. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 45: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.25, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.04 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.02, 95% CI 2-sided [-0.20 to 0.15], Standard Deviation 0.09 — FVC, Day 56. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 46: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.18, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.06 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.02, 95% CI 2-sided [-0.20 to 0.15], Standard Deviation 0.09 — FVC, Day 56. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 47: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.12, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.08 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.02, 95% CI 2-sided [-0.20 to 0.15], Standard Deviation 0.09 — FVC, Day 56. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 48: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.07, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.10 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.02, 95% CI 2-sided [-0.20 to 0.15], Standard Deviation 0.09 — FVC, Day 56. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 49: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.45, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.01, 95% CI 2-sided [-0.20 to 0.17], Standard Deviation 0.10 — FVC, Day 112. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 50: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.37, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.02 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.01, 95% CI 2-sided [-0.20 to 0.17], Standard Deviation 0.10 — FVC, Day 112. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 51: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.30, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.04 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.01, 95% CI 2-sided [-0.20 to 0.17], Standard Deviation 0.10 — FVC, Day 112. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 52: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.22, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.06 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.01, 95% CI 2-sided [-0.20 to 0.17], Standard Deviation 0.10 — FVC, Day 112. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 53: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.17, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.08 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.01, 95% CI 2-sided [-0.20 to 0.17], Standard Deviation 0.10 — FVC, Day 112. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 54: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.12, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.10 L is presented; P-value is actually a posterior probability; Posterior mean difference = -0.01, 95% CI 2-sided [-0.20 to 0.17], Standard Deviation 0.10 — FVC, Day 112. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 55: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.72, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.05, 95% CI 2-sided [-0.13 to 0.24], Standard Deviation 0.09 — FVC, Day 168. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 56: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.65, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.02 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.05, 95% CI 2-sided [-0.13 to 0.24], Standard Deviation 0.09 — FVC, Day 168. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 57: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.57, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.04 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.05, 95% CI 2-sided [-0.13 to 0.24], Standard Deviation 0.09 — FVC, Day 168. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 58: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.48, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.06 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.05, 95% CI 2-sided [-0.13 to 0.24], Standard Deviation 0.09 — FVC, Day 168. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 59: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.39, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.08 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.05, 95% CI 2-sided [-0.13 to 0.24], Standard Deviation 0.09 — FVC, Day 168. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 60: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.30, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.10 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.05, 95% CI 2-sided [-0.13 to 0.24], Standard Deviation 0.09 — FVC, Day 168. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 61: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.76, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.09, 95% CI 2-sided [-0.15 to 0.32], Standard Deviation 0.12 — FVC, Day 280. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 62: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.71, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.02 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.09, 95% CI 2-sided [-0.15 to 0.32], Standard Deviation 0.12 — FVC, Day 280. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 63: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.65, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.04 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.09, 95% CI 2-sided [-0.15 to 0.32], Standard Deviation 0.12 — FVC, Day 280. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 64: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.59, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.06 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.09, 95% CI 2-sided [-0.15 to 0.32], Standard Deviation 0.12 — FVC, Day 280. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 65: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.53, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.08 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.09, 95% CI 2-sided [-0.15 to 0.32], Standard Deviation 0.12 — FVC, Day 280. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 66: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.46, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.10 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.09, 95% CI 2-sided [-0.15 to 0.32], Standard Deviation 0.12 — FVC, Day 280. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 67: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.68, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.05, 95% CI 2-sided [-0.15 to 0.28], Standard Deviation 0.11 — FVC, Day 364. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 68: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.61, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.02 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.05, 95% CI 2-sided [-0.15 to 0.28], Standard Deviation 0.11 — FVC, Day 364. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 69: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.55, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.04 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.05, 95% CI 2-sided [-0.15 to 0.28], Standard Deviation 0.11 — FVC, Day 364. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 70: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.46, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.06 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.05, 95% CI 2-sided [-0.15 to 0.28], Standard Deviation 0.11 — FVC, Day 364. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 71: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.40, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.08 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.05, 95% CI 2-sided [-0.15 to 0.28], Standard Deviation 0.11 — FVC, Day 364. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 72: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.33, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is greater than 0.10 L is presented; P-value is actually a posterior probability; Posterior mean difference = 0.05, 95% CI 2-sided [-0.15 to 0.28], Standard Deviation 0.11 — FVC, Day 364. Data presented are for 95% equal-tailed credible intervals

19. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Danirixin in Part A
Description: Cmax of danirixin was derived from the Pharmacokinetics (PK) samples collected at pre-dose and at 0.5, 1, 2, 4, 6, 8, 10 and 12 hour post-dose on Day 1 and Day 14 in Part A. PK analysis of danirixin was conducted by non-compartmental methods. PK Concenteration Population comprised of par. in the ITT Population and who had provided at least one on-treatment blood sample for determination of danirixin concentration.
Time Frame: Pre-dose and at 0.5, 1, 2, 4, 6, 8, 10 and 12 hour post-dose on Day 1 and Day 14 in Part A
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram per milliliter (ng/mL)
Arm/Group | DNX 50 mg
Number analyzed (Participants) | 9
Nanogram per milliliter (ng/mL)
  Day 1 dose | 397.785 [222.166 to 712.229]
  Day 14 dose | 512.576 [350.162 to 750.324]

20. Primary Outcome: Time of Occurrence of Cmax (Tmax) of Danirixin in Part A
Description: Tmax of danirixin was derived from the PK samples collected at pre-dose and at 0.5, 1, 2, 4, 6, 8, 10 and 12 hour post-dose on Day 1 and Day 14 in Part A. PK analysis of danirixin was conducted by non-compartmental methods.
Time Frame: Pre-dose and at 0.5, 1, 2, 4, 6, 8, 10 and 12 hour post-dose on Day 1 and Day 14 in Part A
Population: PK Population
Measure: Median (Full Range); unit: Hour
Arm/Group | DNX 50 mg
Number analyzed (Participants) | 9
Hour
  Day 1 dose | 1.017 [0.98 to 4.00]
  Day 14 dose | 2.000 [0.35 to 4.02]

21. Primary Outcome: Area Under the Blood Concentration-time Curve (AUC) Over Dosing Interval (AUC[0-12]) of Danirixin in Part A
Description: AUC (0-12) of danirixin was derived from the PK samples collected at pre-dose and at 0.5, 1, 2, 4, 6, 8, 10 and 12 hour post-dose on Day 1 and Day 14 in Part A. PK analysis of danirixin was conducted by non-compartmental methods. A Bayesian random effects model was performed adjusting for the trial as a random effect. A non-informative normal prior distribution was used. Point estimates and corresponding 90 percent credible intervals were constructed.
Time Frame: Pre-dose and at 0.5, 1, 2, 4, 6, 8, 10 and 12 hour post-dose on Day 1 and Day 14 in Part A
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Hour*ng/mL
Arm/Group | DNX 50 mg
Number analyzed (Participants) | 9
Hour*ng/mL
  Day 1 dose | 2203.522 [1303.851 to 3723.976]
  Day 14 dose | 2838.526 [1907.863 to 4223.171]

22. Primary Outcome: Number of Health Care Resource Utilization (HCRU) Defined COPD Exacerbations Per Year in Part B
Description: HCRU COPD exacerbations are defined as moderate or severe exacerbations based on requirement of new prescription antibiotics or oral corticosteroids, hospitalization or emergency room visits for management of COPD exacerbation. For par. with less than 364 days on-treatment, the annual exacerbation rate was imputed as the number of recorded on-treatment exacerbations, divided by the number of 4-week treatment period intervals for which the par. was in the study, multiplied by 13. For par. with 364 or more days on-treatment, the annual exacerbation rate was calculated as the number of recorded exacerbations between study days 1 and 364. Statistical analysis was done using a Bayesian Cox model, assuming a negative binomial distribution for the underlying exacerbation rate. The exacerbation rates along with the ratio (danirixin/placebo), were estimated and corresponding 95 percent credible intervals were produced using non-informative priors. 1 par. was excluded from the analysis.
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Exacerbations per year
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 23 | 20
Exacerbations per year | 2.9 (3.13) | 3.2 (5.82)
Statistical Analysis 1: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.013, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 1.0 is presented; P-value is actually a posterior probability; Posterior mean difference = 2.48, 95% CI 2-sided [0.92 to 4.43], Standard Deviation 0.977 — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 2: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.006, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0.9 is presented; P-value is actually a posterior probability; Posterior mean difference = 2.48, 95% CI 2-sided [0.92 to 4.43], Standard Deviation 0.977 — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 3: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.003, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0.8 is presented; P-value is actually a posterior probability; Posterior mean difference = 2.48, 95% CI 2-sided [0.92 to 4.43], Standard Deviation 0.977 — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 4: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.001, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = 2.48, 95% CI 2-sided [0.92 to 4.43], Standard Deviation 0.977 — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 5: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p < 0.001, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0.6 is presented; P-value is actually a posterior probability; Posterior mean difference = 2.48, 95% CI 2-sided [0.92 to 4.43], Standard Deviation 0.977 — Data presented are for 95% equal-tailed credible intervals

23. Primary Outcome: Monthly Weighted Means of Exacerbations of Chronic Pulmonary Disease Tool-respiratory Symptoms (EXACT-RS) Total Score in Part B
Description: EXACT-RS is a tool which consists of 11 items from the 14 item EXACT- patient reported outcomes (EXACT-PRO) instrument, intended to capture information related to the respiratory symptoms of COPD, i.e. breathlessness, cough, sputum production, chest congestion and chest tightness. The EXACT-RS has a scoring range of 0-40, higher scores indicate more severe symptoms. A par. had at least 10 days of diary data in any month to contribute a non-missing weighted mean AUC of daily values; otherwise the weighted mean for that month were considered missing. A mixed effects model in a Bayesian framework with repeated measures were performed on the EXACT-RS monthly weighted mean AUC data. The posterior mean and corresponding 95 percent credible interval were calculated. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
Score on a scale
  EXACT-RS, 1 month, n=48,45 | 12.4 (5.86) | 11.8 (5.87)
  EXACT-RS, 2 month, n=47,44 | 12.5 (6.67) | 11.6 (6.31)
  EXACT-RS, 3 month, n=46,41 | 12.5 (7.03) | 10.5 (6.33)
  EXACT-RS, 4 month, n=46,41 | 12.4 (6.97) | 10.6 (6.61)
  EXACT-RS, 5 month, n=46,40 | 12.0 (7.12) | 10.6 (6.65)
  EXACT-RS, 6 month, n=44,39 | 12.4 (7.34) | 10.4 (6.14)
  EXACT-RS, 7 month, n=44,39 | 12.3 (7.16) | 10.3 (6.48)
  EXACT-RS, 8 month, n=43,39 | 12.4 (7.3) | 10.3 (6.93)
  EXACT-RS, 9 month, n=40,38 | 12.2 (6.98) | 10.7 (7.08)
  EXACT-RS, 10 month, n=39,38 | 13.0 (7.14) | 10.3 (7.09)
  EXACT-RS, 11 month, n=39,37 | 12.2 (7.23) | 10.5 (6.91)
  EXACT-RS, 12 month, n=39,37 | 12.5 (7.08) | 10.5 (7.12)
Statistical Analysis 1: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.60, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.36, 95% CI 2-sided [-2.81 to 2.17], Standard Deviation 1.29 — EXACT-RS, 1 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 2: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.65, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.58, 95% CI 2-sided [-3.11 to 2.37], Standard Deviation 1.42 — EXACT-RS, 2 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 3: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.83, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.46, 95% CI 2-sided [-4.43 to 1.45], Standard Deviation 1.52 — EXACT-RS, 3 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 4: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.78, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.20, 95% CI 2-sided [-4.07 to 1.90], Standard Deviation 1.53 — EXACT-RS, 4 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 5: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.73, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.96, 95% CI 2-sided [-3.82 to 2.28], Standard Deviation 1.56 — EXACT-RS, 5 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 6: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.72, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.93, 95% CI 2-sided [-4.01 to 2.26], Standard Deviation 1.58 — EXACT-RS, 6 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 7: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.73, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.00, 95% CI 2-sided [-4.15 to 2.09], Standard Deviation 1.58 — EXACT-RS, 7 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 8: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.81, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.48, 95% CI 2-sided [-4.71 to 1.76], Standard Deviation 1.69 — EXACT-RS, 8 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 9: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.76, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.23, 95% CI 2-sided [-4.66 to 2.22], Standard Deviation 1.75 — EXACT-RS, 9 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 10: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.91, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -2.26, 95% CI 2-sided [-5.66 to 0.99], Standard Deviation 1.74 — EXACT-RS, 10 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 11: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.71, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.05, 95% CI 2-sided [-4.73 to 2.13], Standard Deviation 1.73 — EXACT-RS, 11 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 12: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.78, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.35, 95% CI 2-sided [-4.77 to 2.04], Standard Deviation 1.74 — EXACT-RS, 12 month. Data presented are for 95% equal-tailed credible intervals

24. Secondary Outcome: Cmax of Danirixin in Part B
Description: Cmax of danirixin was derived from the PK samples collected at pre-dose and at 0.5, 1, 2, 4, 6, 8, 10 and 12 hour post-dose on Day 1 and Day 364; and at pre-dose and 2 hours on Day 28, 56 and 168 in Part B. PK analysis of danirixin was conducted by non-compartmental methods. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Pre-dose and at 0.5, 1, 2, 4, 6, 8, 10 and 12 hour post-dose on Day 1 and Day 364; and at pre-dose and 2 hours on Day 28, 56 and 168 in Part B
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | DNX 75 mg
Number analyzed (Participants) | 45
ng/mL
  Day 1 dose, n=44 | 517.784 [388.207 to 690.612]
  Day 364 dose, n=36 | 756.391 [554.011 to 1032.700]

25. Secondary Outcome: Tmax of Danirixin in Part B
Description: Tmax of danirixin was derived from the PK samples collected at pre-dose and at 0.5, 1, 2, 4, 6, 8, 10 and 12 hour post-dose on Day 1 and Day 364; and at pre-dose and 2 hours on Day 28, 56 and 168 in Part B. PK analysis of danirixin was conducted by non-compartmental methods. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: as for outcome 24
Population: PK Population
Measure: Median (Full Range); unit: Hour
Arm/Group | DNX 75 mg
Number analyzed (Participants) | 45
Hour
  Day 1 dose, n=44 | 2.000 [0.48 to 6.00]
  Day 364 dose, n=36 | 1.100 [0.50 to 10.00]

26. Secondary Outcome: AUC(0-12) of Danirixin in Part B
Description: AUC (0-12) of danirixin was derived from the PK samples collected at pre-dose and at 0.5, 1, 2, 4, 6, 8, 10 and 12 hour post-dose on Day 1 and Day 364; and at pre-dose and 2 hours on Day 28, 56 and 168 in Part B. PK analysis of danirixin was conducted by non-compartmental methods. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: as for outcome 24
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Hour*ng/mL
Arm/Group | DNX 75 mg
Number analyzed (Participants) | 45
Hour*ng/mL
  Day 1 dose, n=44 | 2388.303 [1834.420 to 3109.425]
  Day 364 dose, n=36 | 4366.995 [3254.122 to 5860.458]

27. Secondary Outcome: Number of EXACT-PRO Exacerbations Per Year in Part B
Description: EXACT-PRO is a 14 item patient reported outcome instrument designed to capture information on the occurrence, frequency, severity, and duration of COPD exacerbations. The total score for EXACT-PRO ranges from 0-100, higher scores indicate more severe symptoms. For par. with less than 364 days on-treatment, the annual exacerbation rate was imputed as the number of recorded on-treatment exacerbations, divided by the number of 4-week treatment period intervals for which the par. was in the study, multiplied by 13. For par. with 364 or more days on-treatment, the annual exacerbation rate was calculated as the number of recorded exacerbations between study days 1 and 364. Statistical analysis was done using a Bayesian Cox model, assuming a negative binomial distribution for the underlying exacerbation rate. The exacerbation rates and the ratio (danirixin/placebo), were estimated and 95 percent credible intervals were produced using non-informative priors. 1 par. was excluded from analysis.
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Exacerbations per year
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 27 | 28
Exacerbations per year | 3.6 (2.75) | 3.3 (3.47)
Statistical Analysis 1: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.278, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 1.0 is presented; P-value is actually a posterior probability; Posterior mean difference = 1.15, 95% CI 2-sided [0.71 to 1.63], Standard Deviation 0.242 — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 2: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.138, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0.9 is presented; P-value is actually a posterior probability; Posterior mean difference = 1.15, 95% CI 2-sided [0.71 to 1.63], Standard Deviation 0.242 — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 3: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.05, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0.8 is presented; P-value is actually a posterior probability; Posterior mean difference = 1.15, 95% CI 2-sided [0.71 to 1.63], Standard Deviation 0.242 — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 4: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.011, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = 1.15, 95% CI 2-sided [0.71 to 1.63], Standard Deviation 0.242 — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 5: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.002, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0.6 is presented; P-value is actually a posterior probability; Posterior mean difference = 1.15, 95% CI 2-sided [0.71 to 1.63], Standard Deviation 0.242 — Data presented are for 95% equal-tailed credible intervals

28. Secondary Outcome: Monthly Weighted Means of Exacerbations of EXACT-PRO Total Score in Part B
Description: EXACT-PRO is a 14 item patient reported outcome instrument designed to capture information on the occurrence, frequency, severity, and duration of COPD exacerbations. The total score for EXACT-PRO ranges from 0-100, higher scores indicate more severe symptoms. A par. had at least 10 days of diary data in any month to contribute a non-missing weighted mean AUC of daily values; otherwise the weighted mean for that month were considered missing. A mixed effects model in a Bayesian framework with repeated measures were performed on the EXACT-PRO monthly weighted mean AUC data. The posterior mean and corresponding 95 percent credible interval were calculated. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
Score on a scale
  EXACT-PRO, 1 month, n=48,45 | 36.5 (9.53) | 35.5 (9.81)
  EXACT-PRO, 2 month, n=47,44 | 36.5 (10.77) | 35.3 (10.69)
  EXACT-PRO, 3 month, n=46,41 | 36.4 (11.23) | 33.6 (10.84)
  EXACT-PRO, 4 month, n=46,41 | 36.4 (11.35) | 33.9 (10.91)
  EXACT-PRO, 5 month, n=46,40 | 35.9 (11.84) | 33.8 (11.28)
  EXACT-PRO, 6 month, n=44,39 | 36.8 (11.58) | 33.8 (10.75)
  EXACT-PRO, 7 month, n=44,39 | 36.5 (11.61) | 33.3 (11.15)
  EXACT-PRO, 8 month, n=43,38 | 36.5 (11.82) | 33.7 (11.73)
  EXACT-PRO, 9 month, n=40,36 | 36.3 (11.25) | 35.2 (11.22)
  EXACT-PRO, 10 month, n=39,37 | 37.4 (11.71) | 33.7 (12.20)
  EXACT-PRO, 11 month, n=39,36 | 36.0 (11.87) | 34.6 (11.49)
  EXACT-PRO, 12 month, n=39,35 | 36.7 (11.57) | 35.0 (11.28)
Statistical Analysis 1: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.62, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.57, 95% CI 2-sided [-4.55 to 3.23], Standard Deviation 2.04 — EXACT-PRO, 1 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 2: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.64, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.72, 95% CI 2-sided [-5.03 to 3.60], Standard Deviation 2.21 — EXACT-PRO, 2 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 3: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.81, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.99, 95% CI 2-sided [-6.60 to 2.27], Standard Deviation 2.29 — EXACT-PRO, 3 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 4: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.77, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.64, 95% CI 2-sided [-5.92 to 3.07], Standard Deviation 2.31 — EXACT-PRO, 4 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 5: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.71, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.30, 95% CI 2-sided [-5.70 to 3.55], Standard Deviation 2.40 — EXACT-PRO, 5 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 6: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.70, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.31, 95% CI 2-sided [-6.46 to 3.05], Standard Deviation 2.42 — EXACT-PRO, 6 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 7: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.74, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.60, 95% CI 2-sided [-6.75 to 2.90], Standard Deviation 2.45 — EXACT-PRO, 7 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 8: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.79, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -2.10, 95% CI 2-sided [-6.93 to 3.30], Standard Deviation 2.63 — EXACT-PRO, 8 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 9: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.77, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.92, 95% CI 2-sided [-7.04 to 3.18], Standard Deviation 2.63 — EXACT-PRO, 9 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 10: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.90, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -3.44, 95% CI 2-sided [-8.74 to 1.87], Standard Deviation 2.72 — EXACT-PRO, 10 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 11: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.66, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.16, 95% CI 2-sided [-6.20 to 4.20], Standard Deviation 2.72 — EXACT-PRO, 11 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 12: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.74, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.73, 95% CI 2-sided [-6.91 to 3.45], Standard Deviation 2.70 — EXACT-PRO, 12 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 13: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.43, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.57, 95% CI 2-sided [-4.55 to 3.23], Standard Deviation 2.04 — EXACT-PRO, 1 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 14: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.45, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.72, 95% CI 2-sided [-5.03 to 3.60], Standard Deviation 2.21 — EXACT-PRO, 2 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 15: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.67, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.99, 95% CI 2-sided [-6.60 to 2.27], Standard Deviation 2.29 — EXACT-PRO, 3 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 16: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.62, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.64, 95% CI 2-sided [-5.92 to 3.07], Standard Deviation 2.31 — EXACT-PRO, 4 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 17: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.55, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.30, 95% CI 2-sided [-5.70 to 3.55], Standard Deviation 2.40 — EXACT-PRO, 5 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 18: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.55, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.31, 95% CI 2-sided [-6.46 to 3.05], Standard Deviation 2.42 — EXACT-PRO, 6 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 19: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.59, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.60, 95% CI 2-sided [-6.75 to 2.90], Standard Deviation 2.45 — EXACT-PRO, 7 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 20: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.65, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -2.10, 95% CI 2-sided [-6.93 to 3.30], Standard Deviation 2.63 — EXACT-PRO, 8 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 21: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.63, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.92, 95% CI 2-sided [-7.04 to 3.18], Standard Deviation 2.63 — EXACT-PRO, 9 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 22: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.81, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -3.44, 95% CI 2-sided [-8.74 to 1.87], Standard Deviation 2.72 — EXACT-PRO, 10 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 23: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.52, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.16, 95% CI 2-sided [-6.20 to 4.20], Standard Deviation 2.72 — EXACT-PRO, 11 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 24: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.60, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.73, 95% CI 2-sided [-6.91 to 3.45], Standard Deviation 2.70 — EXACT-PRO, 12 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 25: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.24, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -2 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.57, 95% CI 2-sided [-4.55 to 3.23], Standard Deviation 2.04 — EXACT-PRO, 1 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 26: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.28, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -2 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.72, 95% CI 2-sided [-5.03 to 3.60], Standard Deviation 2.21 — EXACT-PRO, 2 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 27: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.50, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -2 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.99, 95% CI 2-sided [-6.60 to 2.27], Standard Deviation 2.29 — EXACT-PRO, 3 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 28: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.43, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -2 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.64, 95% CI 2-sided [-5.92 to 3.07], Standard Deviation 2.31 — EXACT-PRO, 4 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 29: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.37, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -2 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.30, 95% CI 2-sided [-5.70 to 3.55], Standard Deviation 2.40 — EXACT-PRO, 5 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 30: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.38, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -2 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.31, 95% CI 2-sided [-6.46 to 3.05], Standard Deviation 2.42 — EXACT-PRO, 6 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 31: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.43, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -2 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.60, 95% CI 2-sided [-6.75 to 2.90], Standard Deviation 2.45 — EXACT-PRO, 7 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 32: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.51, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -2 is presented; P-value is actually a posterior probability; Posterior mean difference = -2.10, 95% CI 2-sided [-6.93 to 3.30], Standard Deviation 2.63 — EXACT-PRO, 8 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 33: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.50, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -2 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.92, 95% CI 2-sided [-7.04 to 3.18], Standard Deviation 2.63 — EXACT-PRO, 9 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 34: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.70, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -2 is presented; P-value is actually a posterior probability; Posterior mean difference = -3.44, 95% CI 2-sided [-8.74 to 1.87], Standard Deviation 2.72 — EXACT-PRO, 10 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 35: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.38, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -2 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.16, 95% CI 2-sided [-6.20 to 4.20], Standard Deviation 2.72 — EXACT-PRO, 11 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 36: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.45, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -2 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.73, 95% CI 2-sided [-6.91 to 3.45], Standard Deviation 2.70 — EXACT-PRO, 12 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 37: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.11, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -3 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.57, 95% CI 2-sided [-4.55 to 3.23], Standard Deviation 2.04 — EXACT-PRO, 1 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 38: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.15, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -3 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.72, 95% CI 2-sided [-5.03 to 3.60], Standard Deviation 2.21 — EXACT-PRO, 2 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 39: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.32, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -3 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.99, 95% CI 2-sided [-6.60 to 2.27], Standard Deviation 2.29 — EXACT-PRO, 3 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 40: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.28, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -3 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.64, 95% CI 2-sided [-5.92 to 3.07], Standard Deviation 2.31 — EXACT-PRO, 4 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 41: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.23, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -3 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.30, 95% CI 2-sided [-5.70 to 3.55], Standard Deviation 2.40 — EXACT-PRO, 5 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 42: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.24, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -3 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.31, 95% CI 2-sided [-6.46 to 3.05], Standard Deviation 2.42 — EXACT-PRO, 6 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 43: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.29, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -3 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.60, 95% CI 2-sided [-6.75 to 2.90], Standard Deviation 2.45 — EXACT-PRO, 7 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 44: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.36, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -3 is presented; P-value is actually a posterior probability; Posterior mean difference = -2.10, 95% CI 2-sided [-6.93 to 3.30], Standard Deviation 2.63 — EXACT-PRO, 8 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 45: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.35, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -3 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.92, 95% CI 2-sided [-7.04 to 3.18], Standard Deviation 2.63 — EXACT-PRO, 9 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 46: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.57, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -3 is presented; P-value is actually a posterior probability; Posterior mean difference = -3.44, 95% CI 2-sided [-8.74 to 1.87], Standard Deviation 2.72 — EXACT-PRO, 10 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 47: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.25, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -3 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.16, 95% CI 2-sided [-6.20 to 4.20], Standard Deviation 2.72 — EXACT-PRO, 11 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 48: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.32, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -3 is presented; P-value is actually a posterior probability; Posterior mean difference = -1.73, 95% CI 2-sided [-6.91 to 3.45], Standard Deviation 2.70 — EXACT-PRO, 12 month. Data presented are for 95% equal-tailed credible intervals

29. Secondary Outcome: Time to First HCRU COPD Exacerbation in Part B
Description: HCRU COPD exacerbations are defined as moderate or severe exacerbations based on requirement of new prescription antibiotics or oral corticosteroids, hospitalization or emergency room visits for management of COPD exacerbation. The time to the first on-treatment HRCU exacerbation were summarized by treatment group. It was analyzed using a Bayesian Cox proportional hazards model. The hazard ratio for the danirixin vs. placebo comparison, along with 95 percent credible interval, was derived, with terms for treatment group, smoking status and country. Posterior probabilities of the ratio of the percentage of par. with an HCRU exacerbation, adjusted for time to first exacerbation, in the danirixin group relative to the placebo group were calculated. 1 par. was excluded from analysis.
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 23 | 20
Days | 166.3 (97.97) | 172.7 (89.66)
Statistical Analysis 1: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.477, Bayesian analysis — Posterior probability that the treatment ratio (DNX 75 mg/ placebo) is less than 1.0 is presented; P-value is actually a posterior probability; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.55 to 1.82] — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 2: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.343, Bayesian analysis — Posterior probability that the treatment ratio (DNX 75 mg/ placebo) is less than 0.9 is presented; P-value is actually a posterior probability; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.55 to 1.82] — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 3: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.221, Bayesian analysis — Posterior probability that the treatment ratio (DNX 75 mg/ placebo) is less than 0.8 is presented; P-value is actually a posterior probability; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.55 to 1.82] — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 4: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.116, Bayesian analysis — Posterior probability that the treatment ratio (DNX 75 mg/ placebo) is less than 0.7 is presented; P-value is actually a posterior probability; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.55 to 1.82] — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 5: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.052, Bayesian analysis — Posterior probability that the treatment ratio (DNX 75 mg/ placebo) is less than 0.6 is presented; P-value is actually a posterior probability; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.55 to 1.82] — Data presented are for 95% equal-tailed credible intervals

30. Secondary Outcome: Time to First EXACT-PRO Event in Part B
Description: The hazard ratio for the DNX versus placebo comparison, along with 95% credible interval and posterior probability was derived and a Bayesian Cox proportional hazards model was used for statistical analysis. The analysis was performed on ITT Population. One participant was excluded from analysis.
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 27 | 28
Days | 101.0 (100.18) | 114.7 (91.16)
Statistical Analysis 1: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.212, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 1.0 is presented; P-value is actually a posterior probability; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.73 to 2.11] — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 2: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.111, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0.9 is presented; P-value is actually a posterior probability; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.73 to 2.11] — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 3: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.049, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0.8 is presented; P-value is actually a posterior probability; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.73 to 2.11] — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 4: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.012, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0.7 is presented; P-value is actually a posterior probability; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.73 to 2.11] — Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 5: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.001, Bayesian Cox analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0.6 is presented; P-value is actually a posterior probability; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.73 to 2.11] — Data presented are for 95% equal-tailed credible intervals

31. Secondary Outcome: Assessment of Duration of EXACT-PRO Events in Part B
Description: Duration is the length of time in days from onset to recovery. It was calculated as the difference in days between day of onset and day of recovery. Onset of event was identified as either an increase in EXACT-PRO score of >=12 points above the par. current mean Baseline for 2 consecutive days, with Day 1 of the 2 days serving as Day 1 onset of the event, or an increase of >=9 points above the par. current mean Baseline for 3 consecutive days, with Day 1 of the 3 days serving as Day 1 onset of the event. Duration was 3-day rolling average was used, which was initiated on Day 1 of onset and ended on Day 1 of Recovery. Recovery was defined as the first day in which par. experienced a persistent, sustained improvement in their condition i.e. decrease in the rolling average EXACT-PRO total score >=9 point from the maximum observed value (highest rolling average EXACT-PRO total score observed the first 14 days of the event) during the first 14 days of an event that is sustained for 7 days.
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 45 | 48
Days | 33.7 (65.40) | 31.5 (59.27)

32. Secondary Outcome: Assessment of Severity of EXACT-PRO Events in Part B
Description: EXACT-PRO tool was used to measure severity of COPD exacerbations in participants. Severity was indicated by the maximum EXACT-PRO total score during the course of event (from day of onset to day of recovery).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 45 | 48
Score on a scale | 48.8 (13.22) | 49.7 (12.63)

33. Secondary Outcome: Monthly Weighted Means of EXACT-RS Domain Scores in Part B
Description: EXACT-RS is a tool which consists of 11 items from the 14 item EXACT-PRO instrument, intended to capture information related to the respiratory symptoms of COPD. EXACT-RS domains included breathlessness, cough and chest symptoms. The EXACT-RS has a scoring range of 0-40, higher scores indicate more severe symptoms. A par. had at least 10 days of diary data in any month to contribute a non-missing weighted mean AUC of daily values; otherwise the weighted mean for that month were considered missing. A mixed effects model in a Bayesian framework with repeated measures were performed. The posterior mean and corresponding 95 percent credible interval were calculated. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
Score on a scale
  EXACT-RS-breath, 1 month, n=48,45 | 6.0 (3.40) | 5.5 (3.59)
  EXACT-RS-breath, 2 month, n=47,44 | 6.3 (3.77) | 5.5 (3.83)
  EXACT-RS-breath, 3 month, n=46,41 | 6.0 (3.79) | 5.0 (3.75)
  EXACT-RS-breath, 4 month, n=46,41 | 6.0 (3.91) | 5.0 (3.86)
  EXACT-RS-breath, 5 month, n=46,40 | 5.8 (4.05) | 5.0 (3.94)
  EXACT-RS-breath, 6 month, n=44,39 | 6.0 (4.11) | 4.8 (3.73)
  EXACT-RS-breath, 7 month, n=44,39 | 5.9 (4.17) | 4.6 (3.83)
  EXACT-RS-breath, 8 month, n=43,39 | 5.9 (3.93) | 4.9 (3.91)
  EXACT-RS-breath, 9 month, n=40,38 | 5.8 (3.87) | 5.1 (4.05)
  EXACT-RS-breath, 10 month, n=39,38 | 6.1 (3.95) | 4.8 (4.12)
  EXACT-RS-breath, 11 month, n=39,37 | 5.8 (3.96) | 5.0 (4.15)
  EXACT-RS-breath, 12 month, n=39,37 | 5.9 (3.90) | 4.9 (4.19)
  EXACT-RS-chest, 1 month, n=48,45 | 2.6 (1.69) | 2.5 (1.59)
  EXACT-RS-chest, 2 month, n=47,44 | 2.7 (1.94) | 2.4 (1.76)
  EXACT-RS-chest, 3 month, n=46,41 | 2.9 (2.13) | 2.2 (1.85)
  EXACT-RS-chest, 4 month, n=46,41 | 2.8 (2.04) | 2.3 (1.90)
  EXACT-RS-chest, 5 month, n=46,40 | 2.8 (2.08) | 2.3 (1.87)
  EXACT-RS-chest, 6 month, n=44,39 | 2.9 (2.20) | 2.3 (1.67)
  EXACT-RS-chest, 7 month, n=44,39 | 2.8 (2.16) | 2.2 (1.74)
  EXACT-RS-chest, 8 month, n=43,39 | 2.9 (2.27) | 2.3 (1.91)
  EXACT-RS-chest, 9 month, n=40,38 | 2.9 (2.23) | 2.4 (1.87)
  EXACT-RS-chest, 10 month, n=39,38 | 3.1 (2.21) | 2.2 (1.86)
  EXACT-RS-chest, 11 month, n=39,37 | 3.0 (2.35) | 2.3 (1.78)
  EXACT-RS-chest, 12 month, n=39,37 | 3.0 (2.31) | 2.4 (1.83)
  EXACT-RS-cough, 1 month, n=48,45 | 3.8 (1.50) | 3.8 (1.32)
  EXACT-RS-cough, 2 month, n=47,44 | 3.5 (1.80) | 3.7 (1.42)
  EXACT-RS-cough, 3 month, n=46,41 | 3.6 (1.87) | 3.3 (1.55)
  EXACT-RS-cough, 4 month, n=46,41 | 3.6 (1.79) | 3.3 (1.57)
  EXACT-RS-cough, 5 month, n=46,40 | 3.4 (1.76) | 3.3 (1.58)
  EXACT-RS-cough, 6 month, n=44,39 | 3.5 (1.76) | 3.4 (1.54)
  EXACT-RS-cough, 7 month, n=44,39 | 3.6 (1.58) | 3.4 (1.72)
  EXACT-RS-cough, 8 month, n=43,39 | 3.6 (1.74) | 3.2 (1.82)
  EXACT-RS-cough, 9 month, n=40,38 | 3.5 (1.72) | 3.3 (1.83)
  EXACT-RS-cough, 10 month, n=39,38 | 3.8 (1.91) | 3.2 (1.82)
  EXACT-RS-cough, 11 month, n=39,37 | 3.5 (1.88) | 3.3 (1.75)
  EXACT-RS-cough, 12 month, n=39,37 | 3.6 (1.91) | 3.2 (1.70)
Statistical Analysis 1: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.64, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.23, 95% CI 2-sided [-1.53 to 1.25], Standard Deviation 0.72 — EXACT-RS-breath, 1 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 2: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.75, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.53, 95% CI 2-sided [-1.91 to 1.10], Standard Deviation 0.78 — EXACT-RS-breath, 2 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 3: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.77, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.60, 95% CI 2-sided [-2.09 to 0.98], Standard Deviation 0.80 — EXACT-RS-breath, 3 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 4: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.74, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.55, 95% CI 2-sided [-2.23 to 0.87], Standard Deviation 0.81 — EXACT-RS-breath, 4 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 5: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.67, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.36, 95% CI 2-sided [-1.88 to 1.27], Standard Deviation 0.83 — EXACT-RS-breath, 5 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 6: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.69, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.43, 95% CI 2-sided [-1.99 to 1.26], Standard Deviation 0.86 — EXACT-RS-breath, 6 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 7: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.72, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.50, 95% CI 2-sided [-2.10 to 1.08], Standard Deviation 0.85 — EXACT-RS-breath, 7 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 8: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.71, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.50, 95% CI 2-sided [-2.11 to 1.14], Standard Deviation 0.87 — EXACT-RS-breath, 8 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 9: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.66, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.34, 95% CI 2-sided [-2.14 to 1.23], Standard Deviation 0.88 — EXACT-RS-breath, 9 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 10: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.84, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.89, 95% CI 2-sided [-2.71 to 0.69], Standard Deviation 0.89 — EXACT-RS-breath, 10 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 11: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.65, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.36, 95% CI 2-sided [-2.15 to 1.41], Standard Deviation 0.91 — EXACT-RS-breath, 11 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 12: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.71, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.49, 95% CI 2-sided [-2.36 to 1.13], Standard Deviation 0.90 — EXACT-RS-breath, 12 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 13: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.13, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.23, 95% CI 2-sided [-1.53 to 1.25], Standard Deviation 0.72 — EXACT-RS-breath, 1 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 14: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.27, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.53, 95% CI 2-sided [-1.91 to 1.10], Standard Deviation 0.78 — EXACT-RS-breath, 2 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 15: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.31, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.60, 95% CI 2-sided [-2.09 to 0.98], Standard Deviation 0.80 — EXACT-RS-breath, 3 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 16: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.29, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.55, 95% CI 2-sided [-2.23 to 0.87], Standard Deviation 0.81 — EXACT-RS-breath, 4 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 17: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.23, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.36, 95% CI 2-sided [-1.88 to 1.27], Standard Deviation 0.83 — EXACT-RS-breath, 5 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 18: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.26, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.43, 95% CI 2-sided [-1.99 to 1.26], Standard Deviation 0.86 — EXACT-RS-breath, 6 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 19: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.28, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.50, 95% CI 2-sided [-2.10 to 1.08], Standard Deviation 0.85 — EXACT-RS-breath, 7 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 20: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.29, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.50, 95% CI 2-sided [-2.11 to 1.14], Standard Deviation 0.87 — EXACT-RS-breath, 8 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 21: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.23, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.34, 95% CI 2-sided [-2.14 to 1.23], Standard Deviation 0.88 — EXACT-RS-breath, 9 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 22: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.45, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.89, 95% CI 2-sided [-2.71 to 0.69], Standard Deviation 0.89 — EXACT-RS-breath, 10 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 23: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.24, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.36, 95% CI 2-sided [-2.15 to 1.41], Standard Deviation 0.91 — EXACT-RS-breath, 11 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 24: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.28, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.49, 95% CI 2-sided [-2.36 to 1.13], Standard Deviation 0.90 — EXACT-RS-breath, 12 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 25: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.26, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.23, 95% CI 2-sided [-1.53 to 1.25], Standard Deviation 0.72 — EXACT-RS-breath, 1 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 26: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.41, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.53, 95% CI 2-sided [-1.91 to 1.10], Standard Deviation 0.78 — EXACT-RS-breath, 2 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 27: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.46, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.60, 95% CI 2-sided [-2.09 to 0.98], Standard Deviation 0.80 — EXACT-RS-breath, 3 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 28: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.43, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.55, 95% CI 2-sided [-2.23 to 0.87], Standard Deviation 0.81 — EXACT-RS-breath, 4 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 29: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.36, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.36, 95% CI 2-sided [-1.88 to 1.27], Standard Deviation 0.83 — EXACT-RS-breath, 5 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 30: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.39, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.43, 95% CI 2-sided [-1.99 to 1.26], Standard Deviation 0.86 — EXACT-RS-breath, 6 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 31: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.42, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.50, 95% CI 2-sided [-2.10 to 1.08], Standard Deviation 0.85 — EXACT-RS-breath, 7 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 32: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.42, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.50, 95% CI 2-sided [-2.11 to 1.14], Standard Deviation 0.87 — EXACT-RS-breath, 8 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 33: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.35, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.34, 95% CI 2-sided [-2.14 to 1.23], Standard Deviation 0.88 — EXACT-RS-breath, 9 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 34: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.58, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.89, 95% CI 2-sided [-2.71 to 0.69], Standard Deviation 0.89 — EXACT-RS-breath, 10 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 35: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.36, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.36, 95% CI 2-sided [-2.15 to 1.41], Standard Deviation 0.91 — EXACT-RS-breath, 11 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 36: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.41, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.49, 95% CI 2-sided [-2.36 to 1.13], Standard Deviation 0.90 — EXACT-RS-breath, 12 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 37: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.66, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.14, 95% CI 2-sided [-0.84 to 0.52], Standard Deviation 0.35 — EXACT-RS-chest, 1 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 38: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.66, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.17, 95% CI 2-sided [-0.94 to 0.55], Standard Deviation 0.39 — EXACT-RS-chest, 2 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 39: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.91, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.56, 95% CI 2-sided [-1.46 to 0.20], Standard Deviation 0.43 — EXACT-RS-chest, 3 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 40: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.79, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.32, 95% CI 2-sided [-1.16 to 0.44], Standard Deviation 0.41 — EXACT-RS-chest, 4 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 41: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.84, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.40, 95% CI 2-sided [-1.24 to 0.41], Standard Deviation 0.42 — EXACT-RS-chest, 5 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 42: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.81, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.39, 95% CI 2-sided [-1.23 to 0.47], Standard Deviation 0.44 — EXACT-RS-chest, 6 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 43: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.76, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.32, 95% CI 2-sided [-1.14 to 0.56], Standard Deviation 0.44 — EXACT-RS-chest, 7 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 44: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.84, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.48, 95% CI 2-sided [-1.43 to 0.43], Standard Deviation 0.48 — EXACT-RS-chest, 8 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 45: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.83, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.46, 95% CI 2-sided [-1.49 to 0.38], Standard Deviation 0.49 — EXACT-RS-chest, 9 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 46: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.94, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.73, 95% CI 2-sided [-1.68 to 0.20], Standard Deviation 0.49 — EXACT-RS-chest, 10 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 47: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.84, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.49, 95% CI 2-sided [-1.45 to 0.48], Standard Deviation 0.50 — EXACT-RS-chest, 11 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 48: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.81, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.43, 95% CI 2-sided [-1.36 to 0.55], Standard Deviation 0.50 — EXACT-RS-chest, 12 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 49: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.01, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.14, 95% CI 2-sided [-0.84 to 0.52], Standard Deviation 0.35 — EXACT-RS-chest, 1 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 50: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.02, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.17, 95% CI 2-sided [-0.94 to 0.55], Standard Deviation 0.39 — EXACT-RS-chest, 2 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 51: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.15, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.56, 95% CI 2-sided [-1.46 to 0.20], Standard Deviation 0.43 — EXACT-RS-chest, 3 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 52: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.05, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.32, 95% CI 2-sided [-1.16 to 0.44], Standard Deviation 0.41 — EXACT-RS-chest, 4 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 53: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.08, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.40, 95% CI 2-sided [-1.24 to 0.41], Standard Deviation 0.42 — EXACT-RS-chest, 5 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 54: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.08, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.39, 95% CI 2-sided [-1.23 to 0.47], Standard Deviation 0.44 — EXACT-RS-chest, 6 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 55: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.06, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.32, 95% CI 2-sided [-1.14 to 0.56], Standard Deviation 0.44 — EXACT-RS-chest, 7 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 56: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.14, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.48, 95% CI 2-sided [-1.43 to 0.43], Standard Deviation 0.48 — EXACT-RS-chest, 8 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 57: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.14, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.46, 95% CI 2-sided [-1.49 to 0.38], Standard Deviation 0.49 — EXACT-RS-chest, 9 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 58: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.29, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.73, 95% CI 2-sided [-1.68 to 0.20], Standard Deviation 0.49 — EXACT-RS-chest, 10 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 59: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.15, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.49, 95% CI 2-sided [-1.45 to 0.48], Standard Deviation 0.50 — EXACT-RS-chest, 11 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 60: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.13, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -1 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.43, 95% CI 2-sided [-1.36 to 0.55], Standard Deviation 0.50 — EXACT-RS-chest, 12 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 61: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.06, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.14, 95% CI 2-sided [-0.84 to 0.52], Standard Deviation 0.35 — EXACT-RS-chest, 1 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 62: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.09, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.17, 95% CI 2-sided [-0.94 to 0.55], Standard Deviation 0.39 — EXACT-RS-chest, 2 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 63: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.37, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.56, 95% CI 2-sided [-1.46 to 0.20], Standard Deviation 0.43 — EXACT-RS-chest, 3 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 64: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.18, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.32, 95% CI 2-sided [-1.16 to 0.44], Standard Deviation 0.41 — EXACT-RS-chest, 4 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 65: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.24, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.40, 95% CI 2-sided [-1.24 to 0.41], Standard Deviation 0.42 — EXACT-RS-chest, 5 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 66: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.24, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.39, 95% CI 2-sided [-1.23 to 0.47], Standard Deviation 0.44 — EXACT-RS-chest, 6 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 67: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.19, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.32, 95% CI 2-sided [-1.14 to 0.56], Standard Deviation 0.44 — EXACT-RS-chest, 7 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 68: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.32, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.48, 95% CI 2-sided [-1.43 to 0.43], Standard Deviation 0.48 — EXACT-RS-chest, 8 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 69: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.32, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.46, 95% CI 2-sided [-1.49 to 0.38], Standard Deviation 0.49 — EXACT-RS-chest, 9 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 70: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.52, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.73, 95% CI 2-sided [-1.68 to 0.20], Standard Deviation 0.49 — EXACT-RS-chest, 10 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 71: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.33, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.49, 95% CI 2-sided [-1.45 to 0.48], Standard Deviation 0.50 — EXACT-RS-chest, 11 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 72: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.29, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.43, 95% CI 2-sided [-1.36 to 0.55], Standard Deviation 0.50 — EXACT-RS-chest, 12 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 73: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.43, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = 0.06, 95% CI 2-sided [-0.59 to 0.62], Standard Deviation 0.31 — EXACT-RS-cough, 1 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 74: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.29, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = 0.19, 95% CI 2-sided [-0.53 to 0.85], Standard Deviation 0.35 — EXACT-RS-cough, 2 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 75: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.70, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.20, 95% CI 2-sided [-0.94 to 0.52], Standard Deviation 0.38 — EXACT-RS-cough, 3 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 76: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.71, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.21, 95% CI 2-sided [-0.92 to 0.50], Standard Deviation 0.37 — EXACT-RS-cough, 4 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 77: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.61, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.11, 95% CI 2-sided [-0.82 to 0.61], Standard Deviation 0.37 — EXACT-RS-cough, 5 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 78: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.48, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = 0.02, 95% CI 2-sided [-0.69 to 0.69], Standard Deviation 0.36 — EXACT-RS-cough, 6 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 79: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.58, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.08, 95% CI 2-sided [-0.79 to 0.62], Standard Deviation 0.36 — EXACT-RS-cough, 7 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 80: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.83, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.39, 95% CI 2-sided [-1.12 to 0.43], Standard Deviation 0.40 — EXACT-RS-cough, 8 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 81: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.74, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.26, 95% CI 2-sided [-1.07 to 0.52], Standard Deviation 0.41 — EXACT-RS-cough, 9 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 82: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.89, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.53, 95% CI 2-sided [-1.40 to 0.29], Standard Deviation 0.43 — EXACT-RS-cough, 10 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 83: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.59, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.10, 95% CI 2-sided [-0.89 to 0.69], Standard Deviation 0.41 — EXACT-RS-cough, 11 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 84: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.77, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than 0 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.30, 95% CI 2-sided [-1.12 to 0.54], Standard Deviation 0.42 — EXACT-RS-cough, 12 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 85: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.01, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = 0.06, 95% CI 2-sided [-0.59 to 0.62], Standard Deviation 0.31 — EXACT-RS-cough, 1 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 86: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.01, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = 0.19, 95% CI 2-sided [-0.53 to 0.85], Standard Deviation 0.35 — EXACT-RS-cough, 2 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 87: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.09, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.20, 95% CI 2-sided [-0.94 to 0.52], Standard Deviation 0.38 — EXACT-RS-cough, 3 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 88: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.09, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.21, 95% CI 2-sided [-0.92 to 0.50], Standard Deviation 0.37 — EXACT-RS-cough, 4 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 89: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.05, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.11, 95% CI 2-sided [-0.82 to 0.61], Standard Deviation 0.37 — EXACT-RS-cough, 5 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 90: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.02, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = 0.02, 95% CI 2-sided [-0.69 to 0.69], Standard Deviation 0.36 — EXACT-RS-cough, 6 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 91: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.04, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.08, 95% CI 2-sided [-0.79 to 0.62], Standard Deviation 0.36 — EXACT-RS-cough, 7 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 92: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.22, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.39, 95% CI 2-sided [-1.12 to 0.43], Standard Deviation 0.40 — EXACT-RS-cough, 8 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 93: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.14, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.26, 95% CI 2-sided [-1.07 to 0.52], Standard Deviation 0.41 — EXACT-RS-cough, 9 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 94: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.36, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.53, 95% CI 2-sided [-1.40 to 0.29], Standard Deviation 0.43 — EXACT-RS-cough, 10 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 95: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.07, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.10, 95% CI 2-sided [-0.89 to 0.69], Standard Deviation 0.41 — EXACT-RS-cough, 11 month. Data presented are for 95% equal-tailed credible intervals
Statistical Analysis 96: Comparison: Placebo vs DNX 75 mg; Test type: Superiority or Other; p = 0.17, Bayesian analysis — Posterior probability that the treatment difference (DNX 75 mg-placebo) is less than -0.7 is presented; P-value is actually a posterior probability; Posterior mean difference = -0.30, 95% CI 2-sided [-1.12 to 0.54], Standard Deviation 0.42 — EXACT-RS-cough, 12 month. Data presented are for 95% equal-tailed credible intervals

34. Secondary Outcome: Change From Baseline for COPD Assessment Test (CAT) at the Indicated Time Points in Part B
Description: The CAT is a validated, 8 item questionnaire which has been developed designed to measure overall COPD-related health status for the initial assessment and longitudinal follow up of par. with COPD. Participants completed each question by rating their experience on a 6 point scale ranging from 0 (no impairment) to 5 (maximum impairment) with a total scoring range of 0 - 40. CAT was assessed at Baseline (Day 1), Day 28, Day 112, Day 168, Day 280 and Day 364 where Baseline was considered as score on Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
Score on a scale
  Day 28; n= 43, 37 | -0.6 (5.19) | -0.7 (7.00)
  Day 112; n= 44, 39 | -0.5 (5.53) | -1.0 (9.50)
  Day 168; n= 43, 37 | -0.8 (5.72) | -1.5 (9.11)
  Day 280; n= 36, 35 | -0.6 (6.02) | -1.2 (9.59)
  Day 364; n= 38, 34 | 0.7 (5.78) | -2.1 (8.77)

35. Secondary Outcome: Number of Participants With Physician's Global Assessment (PGA) Readings in Part B
Description: The PGA is a single item clinician reported outcome measure assessing the overall severity of COPD. Physicians rated disease severity on a four point scale ranging from 1-4 (1=mild, 2=moderate, 3=severe, 4=very severe) at Week 0, 4, 8, 16, 24, 40 and 52. Baseline was considered as score on Day 1. A categorical summary of PGA is presented by treatment and visit.Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
Participants
  Baseline; mild; n= 47, 43 | 5 | 2
  Baseline; moderate; n= 47, 43 | 35 | 37
  Baseline; severe; n= 47, 43 | 7 | 4
  Baseline; very severe; n= 47, 43 | 0 | 0
  Week 4; mild; n= 44, 39 | 10 | 8
  Week 4; moderate; n= 44, 39 | 28 | 27
  Week 4; severe; n= 44, 39 | 6 | 3
  Week 4; very severe; n= 44, 39 | 0 | 1
  Week 8; mild; n= 44, 40 | 10 | 8
  Week 8; moderate; n= 44, 40 | 31 | 30
  Week 8; severe; n= 44, 40 | 3 | 2
  Week 8; very severe; n= 44, 40 | 0 | 0
  Week 16; mild; n= 46, 40 | 12 | 6
  Week 16; moderate; n= 46, 40 | 29 | 32
  Week 16; severe; n= 46, 40 | 5 | 2
  Week 16; very severe; n= 46, 40 | 0 | 0
  Week 24; mild; n= 44, 38 | 8 | 9
  Week 24; moderate; n= 44, 38 | 32 | 25
  Week 24; severe; n= 44, 38 | 4 | 4
  Week 24; very severe; n= 44, 38 | 0 | 0
  Week 40; mild; n= 37, 36 | 4 | 6
  Week 40; moderate; n= 37, 36 | 30 | 28
  Week 40; severe; n= 37, 36 | 3 | 2
  Week 40; very severe; n= 37, 36 | 0 | 0
  Week 52; mild; n= 39, 36 | 7 | 11
  Week 52; n= moderate; n= 39, 36 | 28 | 24
  Week 52; severe; n= 39, 36 | 4 | 1
  Week 52; very severe; n= 39, 36 | 0 | 0

36. Secondary Outcome: Number of Participants With Patient Global Rating of Severity (PGRS) Score in Part B
Description: PGRS is a single global question and was asked to participants to rate their COPD severity on a four point scale ranging from 1-4 (1=mild, 2=moderate, 3=severe, 4=very severe). Participants completed PGRS at Week 0, 4, 8, 16, 24, 40 and 52. Baseline was considered as score on Day 1. A categorical summary of PGRS is presented by treatment and visit.Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
Participants
  Baseline; mild; n= 47, 43 | 10 | 6
  Baseline; moderate; n= 47, 43 | 21 | 29
  Baseline; severe; n= 47, 43 | 15 | 8
  Baseline; very severe; n= 47, 43 | 1 | 0
  Week 4; mild; n= 44, 39 | 7 | 7
  Week 4; moderate; n= 44, 39 | 27 | 27
  Week 4; severe; n= 44, 39 | 10 | 4
  Week 4; very severe; n= 44, 39 | 0 | 1
  Week 8; mild; n= 44, 40 | 4 | 7
  Week 8; moderate; n= 44, 40 | 32 | 29
  Week 8; severe; n= 44, 40 | 7 | 4
  Week 8; very severe; n= 44, 40 | 1 | 0
  Week 16; mild; n= 45, 40 | 6 | 8
  Week 16; moderate; n= 45, 40 | 28 | 26
  Week 16; severe; n= 45, 40 | 11 | 6
  Week 16; very severe; n= 45, 40 | 0 | 0
  Week 24; mild; n= 44, 38 | 6 | 9
  Week 24; moderate; n= 44, 38 | 31 | 23
  Week 24; severe; n= 44, 38 | 7 | 6
  Week 24; very severe; n= 44, 38 | 0 | 0
  Week 40; mild; n= 37, 36 | 7 | 9
  Week 40; moderate; n= 37, 36 | 21 | 21
  Week 40; severe; n= 37, 36 | 9 | 6
  Week 40; very severe; n= 37, 36 | 0 | 0
  Week 52; mild; n= 39, 36 | 6 | 7
  Week 52; n= moderate; n= 39, 36 | 24 | 23
  Week 52; severe; n= 39, 36 | 9 | 6
  Week 52; very severe; n= 39, 36 | 0 | 0

37. Secondary Outcome: Number of Participants With Patient Global Impression of Change (PGIC)Score in Part B
Description: Participants completed a PGIC questions at Week 4, 8, 16, 24, 40 and 52. Response options were on a 7 point Likert scale ranging from much better to much worse. PGIC was re-coded from a categorical to numerical value prior to analysis as: much worse = -3, worse = -2, slightly worse = -1, no change = 0, slightly better = 1, better = 2, much better = 3.A categorical summary of PGIC is presented by treatment and visit.Only those participants with data available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Up to Day 392 in Part B
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | DNX 75 mg
Number analyzed (Participants) | 48 | 45
Participants
  Week 4; much worse; n= 44, 39 | 0 | 1
  Week 4; worse; n= 44, 39 | 1 | 4
  Week 4; slightly worse; n= 44, 39 | 1 | 0
  Week 4; no change; n= 44, 39 | 18 | 17
  Week 4; slightly better; n= 44, 39 | 15 | 12
  Week 4; better; n= 44, 39 | 9 | 4
  Week 4; much better; n= 44, 39 | 0 | 1
  Week 8; much worse; n= 44, 39 | 1 | 0
  Week 8; worse; n= 44, 39 | 1 | 1
  Week 8; slightly worse; n= 44, 39 | 6 | 5
  Week 8; no change; n= 44, 39 | 16 | 18
  Week 8; slightly better; n= 44, 39 | 15 | 10
  Week 8; better; n= 44, 39 | 4 | 4
  Week 8; much better; n= 44, 39 | 1 | 1
  Week 16; much worse; n= 45, 40 | 0 | 1
  Week 16; worse; n= 45, 40 | 0 | 1
  Week 16; slightly worse; n= 45, 40 | 0 | 3
  Week 16; no change; n= 45, 40 | 21 | 17
  Week 16; slightly better; n= 45, 40 | 20 | 13
  Week 16; better; n= 45, 40 | 3 | 2
  Week 16; much better; n= 45, 40 | 1 | 3
  Week 24; much worse; n= 44, 38 | 0 | 1
  Week 4; worse; n= 44, 38 | 1 | 2
  Week 24; slightly worse; n= 44, 38 | 3 | 3
  Week 24; no change; n= 44, 38 | 15 | 13
  Week 24; slightly better; n= 44, 38 | 16 | 9
  Week 24; better; n= 44, 38 | 8 | 8
  Week 24; much better; n= 44, 38 | 1 | 2
  Week 40; much worse; n= 37, 36 | 0 | 0
  Week 40; worse; n= 37, 36 | 2 | 1
  Week 40; slightly worse; n= 37, 36 | 3 | 7
  Week 40; no change; n=37, 36 | 9 | 12
  Week 40; slightly better; n=37, 36 | 14 | 7
  Week 40; better; n= 37, 36 | 7 | 7
  Week 40; much better; n= 37, 36 | 2 | 2
  Week 52; much worse; n= 39, 35 | 0 | 1
  Week 52; worse; n= 39, 35 | 1 | 0
  Week 52; slightly worse; n= 39, 35 | 3 | 7
  Week 52; no change; n= 39, 35 | 14 | 15
  Week 52; slightly better; n= 39, 35 | 9 | 4
  Week 52; better; n= 39, 35 | 11 | 5
  Week 52; much better; n= 39, 35 | 1 | 3

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study treatment up to Day 28 in Part A and up to Day 392 in Part B.
Description: On treatment SAEs and non-serious AEs were reported for the All Subjects Population.
Arm/Group | DNX 50 mg | Placebo | DNX 75 mg
Serious Adverse Events (participants affected / at risk) | 1/9 | 10/48 | 10/45
Other Adverse Events (participants affected / at risk) | 5/9 | 25/48 | 25/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DNX 50 mg (N=9) | Placebo (N=48) | DNX 75 mg (N=45)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1
Cholangitis sclerosing (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 0
Cholangitis infective (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gallbladder adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 1
Brain injury (Nervous system disorders) | 0 | 1 | 0
Device loosening (Product Issues) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DNX 50 mg (N=9) | Placebo (N=48) | DNX 75 mg (N=45)
Nausea (Gastrointestinal disorders) | 1 | 2 | 0
Fatigue (General disorders) | 1 | 0 | 3
Malaise (General disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 16 | 13
Headache (Nervous system disorders) | 1 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hyperhidrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 0
Diarrhoea (General disorders) | 0 | 8 | 4
Cystitis (Infections and infestations) | 0 | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.